CLINICAL TRIAL: NCT04156074
Title: Innovative Food Structures to Enhance the Sensory Experience, the Nutrient Profile and Nutrient Bioavailability for Older People
Brief Title: Innovative Food Structures to Enhance Nutrient Bioavailability
Acronym: NutriPlus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Collaborators: Department of Agriculture Food and the Marine (Unknown)
Responsible Party: Principal Investigator, Aifric O'Sullivan, Assistant Professor, University College Dublin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LS-19-56-McCourt-OSullivan
Record Dates: First submitted 2019-11-05; First posted 2019-11-07 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Vitamin D Deficiency; Aging Well
Keywords: Vitamin D; Bioavailability; Aging; Fortified foods; Vitamin D status; 25-hydroxyvitamin D
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Intervention Model Description: Parallel Randomized Controlled Trial
Who Masked: Participant, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Vitamin D enriched (20 mcg/day) olive oil emulsion drink (Experimental): 30 mL vitamin D enriched drink consumed daily for 4 weeks
  Interventions: Dietary Supplement: Vitamin D enriched (20 mcg/day) olive oil emulsion drink
- Vitamin D enriched (20 mcg/day) coconut oil emulsion drink (Active Comparator): 30 mL vitamin D enriched drink consumed daily for 4 weeks
  Interventions: Dietary Supplement: Vitamin D enriched (20 mcg/day) coconut oil emulsion drink
- Placebo coconut oil emulsion drink (Placebo Comparator): 30 mL placebo drink consumed daily for 4 weeks
  Interventions: Dietary Supplement: Placebo coconut oil emulsion drink
- Vitamin D supplement (20 mcg/day) (Active Comparator): Vitamin D supplement consumed daily for 4 weeks
  Interventions: Dietary Supplement: Vitamin D supplement (20 mcg/day)

INTERVENTIONS:
Dietary Supplement: Vitamin D enriched (20 mcg/day) olive oil emulsion drink — Vitamin D enriched (20 mcg/day) olive oil emulsion drink. 30 mL drink daily
  Arms: Vitamin D enriched (20 mcg/day) olive oil emulsion drink
Dietary Supplement: Vitamin D enriched (20 mcg/day) coconut oil emulsion drink — Vitamin D enriched (20 mcg/day) coconut oil emulsion drink 30 mL drink daily
  Arms: Vitamin D enriched (20 mcg/day) coconut oil emulsion drink
Dietary Supplement: Placebo coconut oil emulsion drink — Placebo coconut oil emulsion drink 30 mL drink daily
  Arms: Placebo coconut oil emulsion drink
Dietary Supplement: Vitamin D supplement (20 mcg/day) — Vitamin D supplement (20 mcg/day) Pill consumed daily
  Arms: Vitamin D supplement (20 mcg/day)

SUMMARY:
This randomized controlled trial (RCT) will compare the change in vitamin D status (25-hydroxyvitamin D nmol/L) after a 4 week intervention with 4 groups:

1. Vitamin D enriched (20ug) olive oil emulsion drink
2. Vitamin D enriched (20ug) coconut oil emulsion drink
3. Placebo emulsion drink
4. Vitamin D supplement (20ug) Participants will be randomized to 1 of 4 intervention group.

Hypothesis 1: 25-hydroxyvitamin D concentrations are higher in the olive oil emulsion drink group compared to the placebo emulsion drink group post intervention.

Hypothesis 2: 25-hydroxyvitamin D concentrations are higher in the olive oil emulsion drink group compared to the coconut oil emulsion drink group post intervention.

ELIGIBILITY:
Inclusion Criteria:

• Healthy adults

Exclusion Criteria:

* Pregnant/lactating
* Smokers
* Individuals who are not free-living
* An inability to read, write or understand English
* Following a strict diet for any reason, insulin dependent diabetes, coeliac etc.
* Disease that requires chronic therapeutic nutritional or medical treatment
* Those with conditions that may affect kidney function
* Those with osteoporosis
* Those taking supplemental vitamin D
* Those who have been on a sun holiday in the last 2 months
* Those with a milk protein allergy or lactose intolerance

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Vitamin D status | Baseline to 28 days
  Change in vitamin D status measured as serum 25-hydroxyvitamin D (nmol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Aifric O'Sullivan, PhD, Principal Investigator — University College Dublin
Locations (1):
- University College Dublin, Dublin, Ireland